CLINICAL TRIAL: NCT04963348
Title: Investigate the Potential of Deep Learning in Assessing Pneumoconiosis Depicted on Digital Chest Radiographs and to Compare Its Performance With Certified Radiologists
Brief Title: Potential of Deep Learning in Assessing Pneumoconiosis Depicted on Digital Chest Radiography
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019467
Record Dates: First submitted 2021-06-28; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Pneumoconiosis
MeSH Terms: conditions — Pneumoconiosis | interventions — Convolutional Neural Networks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- convolutional neural network (CNN): a classical deep convolutional neural network (CNN) called Inception-V3 was applied to the image sets and validated the classification performance of the trained models
  Interventions: Other: convolutional neural networks (CNNs)

INTERVENTIONS:
Other: convolutional neural networks (CNNs) — CNN architecture named U-Net architecture
  Other Names: deep learning technology

SUMMARY:
Pneumoconiosis is relatively prevalent in low/middle-income countries, and it remains a challenging task to accurately and reliably diagnose pneumoconiosis. The investigators implemented a deep learning solution and clarified the potential of deep learning in pneumoconiosis diagnosis by comparing its performance with two certified radiologists. The deep learning demonstrated a unique potential in classifying pneumoconiosis.

DETAILED DESCRIPTION:
The investigators retrospectively collected a dataset consisting of 1881 chest X-ray images in the form of digital radiography. These images were acquired in a screening setting on subjects who had a history of working in an environment that exposed them to harmful dust. Among these subjects, 923 were diagnosed with pneumoconiosis, and 958 were normal. To identify the subjects with pneumoconiosis, the investigators applied a classical deep convolutional neural network (CNN) called Inception-V3 to these image sets and validated the classification performance of the trained models using the area under the receiver operating characteristic curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* industrial workers with a history of exposure to dust and underwent DR screening of pneumoconiosis from 2015 to 2018

Exclusion Criteria:

* patients with poor image quality
* patients with incomplete clinical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Of these subjects, 923 were diagnosed with pneumoconiosis, 958 were normal. Among these subjects, 163 were females.
Sampling Method: Non-Probability Sample
Enrollment: 1881 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
the diagnosis of pneumoconiosis | up to 6 months
  The diagnosis and staging of pneumoconiosis were made by an expert panel consisting of certified radiologists and occupational physicians. The diagnosis of pneumoconiosis was confirmed by medical history and previous medical records(chest X-rays and pulmonary function testing).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wang, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No